CLINICAL TRIAL: NCT05494125
Title: Effects of Continuous Erector Spinae Plane Blocks on Recovery, Pain and Opioid Consumption After Multilevel Spine Surgery: A Prospective Randomized Clinical Trial
Brief Title: Effects of Continuous ESP Catheters on Recovery, Pain and Opioid Consumption After Multilevel Spine Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanticipated adverse events occurred in 2 participants
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-1815
Record Dates: First submitted 2022-07-15; First posted 2022-08-09 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain; Spine Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Catheters with Ropivacaine 0.2% (Experimental)
  Interventions: Other: Ropivacaine
- ESP Catheters with Saline Solution (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ropivacaine — Patients will receive a continuous infusion of ropivacaine through bilateral ESP catheters
  Arms: ESP Catheters with Ropivacaine 0.2%
Other: Placebo — Patients will receive a continuous infusion of saline solution through bilateral ESP catheters
  Arms: ESP Catheters with Saline Solution

SUMMARY:
Single-shot erector spinae plane (ESP) blocks (ESPB) are emerging as an intervention to improve pain and minimize opioid consumption after lumbar spine surgery. Although promising, there is minimal evidence to support routine use, and widespread clinical adoption may be limited to centers with advanced regional anesthesia resources and expertise. Continuous ESP catheter techniques may solve these problems but are associated with challenges of their own. This trial will investigate the role of adding surgeon-placed, continuous ESP catheters to single-shot ESPBs for patients undergoing multilevel spine surgery. It will assess whether adding ESP catheters with ropivacaine infusion for 48 hours after surgery offers opioid-minimizing analgesia and improves patient quality of recovery, compared to ESP catheters with saline/placebo infusion for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Presenting for elective multilevel (>2 spinal levels) spinal fusion
* Lumbar, thoracic, and thoracolumbar procedures included
* Posterior surgical approach
* Willing and able to follow the study protocol
* Able to provide informed consent

Exclusion Criteria:

* Opioid tolerance (more than 60 morphine milliequivalents daily for more than 3 months)
* Daily gabapentin/pregabalin use for longer than 3 months
* Prior spine surgery at the index level
* Allergy or contraindication (including renal, liver disease) to included study medications
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Number of patients who require escalation to (ie, a new prescription for) an opioid-iv-patient controlled analgesia (iv-PCA) | First 72 hours after surgery

SECONDARY OUTCOMES:
Duration of use and dose of opioid-iv-pca (if required) | First 72 hours after surgery
  Measured in morphine equivalents daily
Post-operative opioid consumption | From PACU arrival to 72 hours post surgery
  Measured in morphine equivalents daily
Numeric rating scale (NRS) pain scores: every 8 hours | Between PACU and 72 hours post surgery
  Scale of 0-10, 0 being no pain, 10 being the worst pain possible
Quality of Recovery 15 (QoR15) scores | Pre-operative, holding area/day of surgery, 24 hours, 48 hours, 14 days and 42 days post surgery
  The Quality of Recovery 15 (QoR15) is a 15-item questionnaire which assesses five domains of patient-reported health status: pain, physical comfort, physical independence, psychological support and emotional state. It has a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).
Duration of ESP catheter(s) use and reasons (if any) for catheter failure or dislodgement | First 48 hours post surgery
  Measured in days after placement
Total dose of ropivacaine delivered | First 48 hours post surgery
  Measured in mg/kg/hr
Opioid-related side effects (nausea, vomiting, anti-emetic medication administration, constipation, sedation, administration of naloxone) | First 48 hours post surgery
  If the patient ever had any of the events
Length of hospital stay | From PACU arrival to hospital discharge, up to 2 weeks
  Measured in days after surgery
Patient satisfaction scale with pain management and ESP catheters | First 72 hours, 14 days, and 42 days post surgery
  Patient satisfaction will be assessed using a 0 to 10 scale (0 being not satisfied to 10 being totally satisfied)
Incidence of ongoing pain and opioid consumption, measured at 3 and 6 months post-surgery | 3 and 6 month post surgery
  Measured with a 7-item questionnaire to assess chronic pain and opioid use

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Amoroso K, Hughes AP, Sama AA, Cammisa FP, Shue J, Soffin EM. Continuous erector spinae plane catheters leading to unwanted neuraxial spread after spinal fusion surgery: a report of two cases from a terminated prospective randomized clinical trial. Reg Anesth Pain Med. 2023 Sep;48(9):478-481. doi: 10.1136/rapm-2023-104587. Epub 2023 May 16. PMID 37192785